CLINICAL TRIAL: NCT03580161
Title: Simplification of Low Level Internal Dosimetry
Acronym: SOLLID
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4767
Record Dates: First submitted 2018-06-21; First posted 2018-07-09 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Exposure to Medical Diagnostic Radiation
Keywords: Absorbed Radiation Dose; Radiation Risks; Radiation Protection; Dosimetry
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 18-F FDG PET/CT: Patients receiving routine diagnostic scan
  Interventions: Other: 18-F FDG PET/CT dosimetry scans and measurements
- Ga-68 PSMA PET/CT: Patients receiving routine diagnostic scan
  Interventions: Other: Ga-68 PSMA PET/CT dosimetry scans and measurements
- 68-Ga Dotatate PET/CT: Patients receiving routine diagnostic scan
  Interventions: Other: 68-Ga Dotatate PET/CT dosimetry scans and measurements
- 99mTc Pertechnetate Thyroid Scan: Patients receiving routine diagnostic scan
  Interventions: Other: 99mTc Pertechnetate Thyroid dosimetry scans and measurements
- 99mTc DMSA(III) Renal Scan: Patients receiving routine diagnostic scan
  Interventions: Other: 99mTc DMSA(III) Renal dosimetry scans and measurements
- 99mTc MAG3 Renal Scan: Patients receiving routine diagnostic scan
  Interventions: Other: 99mTc MAG3 Renal dosimetry scans and measurements
- 99mTc MDP/HDP Bone Scan: Patients receiving routine diagnostic scan
  Interventions: Other: 99mTc MDP/HDP Bone dosimetry scans and measurements

INTERVENTIONS:
Other: 18-F FDG PET/CT dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 18-F FDG PET/CT
Other: Ga-68 PSMA PET/CT dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: Ga-68 PSMA PET/CT
Other: 68-Ga Dotatate PET/CT dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 68-Ga Dotatate PET/CT
Other: 99mTc Pertechnetate Thyroid dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 99mTc Pertechnetate Thyroid Scan
Other: 99mTc DMSA(III) Renal dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 99mTc DMSA(III) Renal Scan
Other: 99mTc MAG3 Renal dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 99mTc MAG3 Renal Scan
Other: 99mTc MDP/HDP Bone dosimetry scans and measurements — Participants will have additional scans and retention measurements for dosimetry alongside their routine diagnostic scans
  Groups: 99mTc MDP/HDP Bone Scan

SUMMARY:
This is a pilot study with the primary aim being to identify the minimum number of scans and measurements necessary to determine accurately the absorbed radiation doses delivered from internal sources of radiation administered for diagnostic nuclear medicine procedures.

DETAILED DESCRIPTION:
A study to develop practical methods of accurate low radiation absorbed dose measurement in patients referred for nuclear medicine scans.

There is currently very little information on and therefore understanding of the effects of exposure to low levels of radiation on patients or radiation workers. Assumptions are largely based on evidence from high radiation doses following nuclear incidents which may not be applicable to medical procedures. Underestimation of the radiation effects incurs greater risk to patients than is currently assumed, while overestimation can prevent more informative scans that would be obtained from higher administered activities. This research study answers an invitation from the Department of Health Policy research programme to improve our understanding of those low radiation dose risks.

Over 600,000 patients have nuclear medicine scans in the UK each year, presenting an opportunity to accurately measure low radiation doses and follow up the effects on a large number of patients. This study will develop practical methods to measure accurately the radiation doses delivered to patients referred for nuclear medicine positron emission tomography (PET) and single photon emission computed tomography (SPECT) scans.

Five patients referred for each of 7 diagnostic nuclear medicine procedures will undergo up to 7 quantitative PET/SPECT scans and up to 10 whole body radiation retention measurements over the course of 1-2 days to enable the absorbed radiation doses to be calculated accurately. Analysis of subsets of these measurements will be performed to identify the timing and minimum number of measurements necessary for accurate dose estimates.

The longer term aim is that these methods and results will subsequently be used to inform a national epidemiological (epidemiology is the study of factors affecting the health and illness of populations) study on the effects of low doses of radiation.

ELIGIBILITY:
Inclusion Criteria:

* All patients able to undergo the procedures necessary to acquire sufficient data for dosimetry, consisting of up 7 nuclear medicine scans and 10 external radiation retention measurements over a time period of up to 24 hours

Exclusion Criteria:

* Patients unable or unwilling to undergo further procedures that may include scans and external retention measurements.
* Paediatric patients 18 years of age and under.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Royal Marsden Hospital patients undergoing diagnostic nuclear medicine procedures to assess bone marrow involvement, kidney function, thyroid function, staging of adult malignancies and glucose metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The uncertainty on the absorbed dose calculation | 6-24 hours
  The uncertainty on the absorbed dose calculation for normal organs and for the whole-body as a function of the number of scans and whole-body counts acquired.

SECONDARY OUTCOMES:
The range of absorbed doses delivered | 6-24 hours
  The range of absorbed doses delivered to healthy organs from 99mTc-MDP/HDP bone imaging, 99mTc- MAG-3 renograms, 99mTc-Pertechnetate thyroid Imaging, 18F-FDG, 68Ga PSMA and 68Ga DOTATATE.

OTHER OUTCOMES:
The range of risk estimates | 6-24 hours
  The range of risk estimates associated with diagnostic procedures, derived from the absorbed doses.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Flux, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flux G, Murray I, Rushforth D, Gape P, Abreu C, Lee M, Ribeiro A, Gregory R, Chittenden S, Thurston J, Du Y, Gear J. SOLLID - a single centre study to develop methods to investigate the effects of low radiation doses within nuclear medicine, to enable multicentre epidemiological investigations. Br J Radiol. 2021 Mar 1;94(1119):20200072. doi: 10.1259/bjr.20200072. Epub 2020 Sep 9. PMID 32903035